CLINICAL TRIAL: NCT07228286
Title: REstoring CONsciousness With NEurostimulation of the Central Thalamus: The RECONNECT Study
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Samuel Snider, MD (Other)
Responsible Party: Sponsor-Investigator, Samuel Snider, MD, Neurointensivist; Assistant Professor of Neurology Harvard Medical School, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Device Feasibility
Other Study IDs: 2025P001898
Record Dates: First submitted 2025-11-07; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Disorders of Consciousness
Keywords: deep brain stimulation; disorders of consciousness; brain injury; thalamus
MeSH Terms: conditions — Consciousness Disorders; Brain Injuries | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- active stimulation (Experimental): Each participant will receive a pre-determined sequence of active stimulation to one of two targets or no stimulation over the course of 10 months. This will be divided into two blocks (each with STIM and OFF periods) targeting each of the two thalamic targets. The order will be reversed in participant 2 relative to participant 1.
  Interventions: Device: Deep brain stimulation (DBS) electrode implantation
- no stimulation (Sham Comparator): periods of no active stimulation intermixed with active stimulation to one of two targets.
  Interventions: Device: Deep brain stimulation (DBS) electrode implantation

INTERVENTIONS:
Device: Deep brain stimulation (DBS) electrode implantation — DBS electrodes implanted to two targets in each thalamus.

SUMMARY:
The RE-CONNECT study is an early feasibility study to establish the safety, feasibility, and efficacy of two central thalamic deep brain stimulation targets in patients with chronic disorders of consciousness.

DETAILED DESCRIPTION:
The overall goal is to collect pilot data on the safety, feasibility, and comparative behavioral efficacy of DBS to two specific thalamic targets in patients with disorders of consciousness (DoC): A sub-region of the centromedian/parafascicular nucleus (CM-Pf) and the centrolateral nucleus (CL). The investigators will recruit 2 participants over two years to participate in a single-center, double-blinded, cross-over study.

After consent, the investigators will first confirm the stability of the clinical DoC diagnosis during a 1-month screening period. The purpose of this phase is to ensure that participants are not already on a trajectory of clinical improvement. Investigators will then implant two DBS electrodes (PerceptTM; Medtronic) into each thalamus, one targeting the thalamic CM-Pf sub-region and the other targeting the CL nucleus. After a one-month recovery period, investigators will titrate stimulation settings, and participants will then enter a 10-month blinded stimulation phase comprising periods of either continuous daily real (STIM-ON) or sham (STIM-OFF) stimulation delivered separately to each target. One participant will receive CM-Pf stimulation blocks first and CL stimulation blocks second; the other participant will receive the reverse target order (CL then CM-Pf). Investigators will enroll two patients, measuring procedure and device-related adverse and serious adverse events, as well as the feasibility of successfully targeting the CM-Pf sub-region. Finally, investigators will measure and compare the magnitude of CM-Pf versus CL stimulation induced changes on a standardized behavioral scale for evaluating patients with DoC.

ELIGIBILITY:
Inclusion Criteria:

* Central nervous system injury of any etiology (e.g., cardiac arrest, traumatic brain injury, ischemic stroke, cerebral hemorrhage, encephalitis) that occurred at least 3 months prior to the eligibility phone call
* The participant does not exhibit either of the following behaviors every day: meaningful interaction (defined as intelligible speech and ability to follow verbal commands) or functional object use
* A CRS-R based diagnosis of DoC; either Unresponsive Wakefulness Syndrome (UWS) or Minimally Conscious State (MCS- or +).
* The participant must have a documented health care proxy or court-appointed guardian
* Neurologist and neurosurgeon consensus review of most recent clinical MRI (if no MRI, then most recent CT) determines there is no bilateral subcortical injury preventing precise placement of electrodes (e.g., major injuries to the bilateral thalami or severe and bilateral subcortical anatomical distortions).

Exclusion Criteria:

* - Pregnant
* Contraindication to brain MRI
* Due to transportation requirements, participants whose primary residence (Skilled Nursing Facility, Long Term Acute Care, or home) is outside the Greater Boston metropolitan area
* Pre-existing psychiatric, neurological or medical condition that makes the patient, in the opinion of the study team, a poor surgical candidate (e.g., neurodegenerative disorder, significant cardiopulmonary disorder, need for chronic anticoagulation)
* Structural abnormality of the chest wall, neck, brain, or skull that makes safe placement of the electrodes, in the opinion of the study team, infeasible or prone to complication
* Neurologist and neurosurgeon consensus review of most recent clinical MRI (if no MRI, then most recent CT) determines there is no bilateral diffuse injury to the basal ganglia
* Medical contraindications to surgery including:

  * Chronic infection
  * Coagulopathy (INR > 1.5, aPTT 45 sec, platelet count < 100 x 103 / uL)
  * Poorly controlled blood pressure (> 2 episodes during screening phase of blood pressure > 180/110 sustained on repeated measurements) and evidence of cardiovascular disease
  * Participation in another drug, device or biological trial within 90 days
  * Current implanted stimulation device (e.g., pacemaker, defibrillator, spinal cord stimulator, deep brain stimulator)
  * Anticoagulant or anti-platelet medication that cannot be safely stopped for > 2.5 weeks in the peri-operative period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Estimated)
Dates: Start 2025-11-10 (Estimated); Primary Completion 2029-02-10 (Estimated); Study Completion 2029-02-10 (Estimated)

PRIMARY OUTCOMES:
Coma Recovery Scale Revised (CRS-R) | Outcomes will be assessed at baseline and weekly during the 12 month study period.
  Behavioral scale for patients wth DoC. Range: 0 to 23 with higher values indicating greater levels of awareness.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided